CLINICAL TRIAL: NCT02450877
Title: A Randomized, Multicenter, Open-label, Phase 2 Study, With a Safety Run-in Part to Evaluate Safety, Pharmacodynamics and Efficacy of Azacitidine Compared to No Anticancer Treatment in Children and Young Adults With Acute Myeloid Leukemia in Molecular Relapse After First Complete Remission
Brief Title: A Study of Safety, Efficacy and Pharmacodynamics of Azacitidine in Children and Young Adults With Acute Myeloid Leukemia.
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Celgene (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: AZA-AML-004
Record Dates: First submitted 2015-05-19; First posted 2015-05-21 (Estimated); Last update posted 2019-12-20 (Actual); Status verified 2019-12

CONDITIONS: Leukemia, Myeloid, Acute
Keywords: Children; Young Adults; Azacitidine; Acute Myeloid Leukemia; Molecular Relapse; Vidaza; AZA-AML-004
MeSH Terms: conditions — Leukemia, Myeloid, Acute | interventions — Azacitidine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Azacitidine Treatment (Experimental): : Subjects randomized to the experimental arm will receive up to 3 cycles of IV azacitidine on Days 1 through 7 at the dose selected from the safety run-in part.
  Interventions: Drug: Azacitidine
- Control Arm: 'Watch and Wait' (Other): Subjects randomized to the control arm will undergo 'watch and wait' until clinical relapse (defined as at least 5% blasts in PB (peripheral blood) and/or BM (bone marrow) and/or proven histological extramedullary relapse).
  Interventions: Other: Control Arm

INTERVENTIONS:
Drug: Azacitidine
  Arms: Azacitidine Treatment
Other: Control Arm
  Arms: Control Arm: 'Watch and Wait'

SUMMARY:
This study is a randomized, multicenter, open-label, Phase 2 study that will be run in 2 parts: a safety run-in part to determine the dose of azacitidine and then a second part to determine the efficacy of that dose in children and young adults with acute myeloid leukemia in molecular relapse after their first complete remission.

Indication Treatment of children and young adults with molecular relapse of acute myeloid leukemia (AML) after first complete remission (CR1).

Objectives Primary Objectives Safety Run-in Part To establish a safe and tolerable dose of azacitidine to be used in the randomized part of the study.

Randomized Part To evaluate the effect of azacitidine treatment in AML subjects at molecular relapse after CR1 when compared to no treatment with regard to the progression-free rate (PFR) at Day 84 (±4 days) post randomization.

Secondary Objectives Safety Run-in Part To establish azacitidine plasma pharmacokinetic (PK) parameters in subjects with molecular relapse AML after CR1 and to assess efficacy.

Randomized Part To evaluate the safety, pharmacodynamics (PD), and efficacy of azacitidine treatment in subjects with molecular relapse AML after CR1.

Study Design The population of this trial consists of children and young adults with AML who achieved a complete response (CR) with molecular remission, defined as Minimal Residual Disease (MRD) less than 5 x 10-4, following their initial induction therapy and who subsequently have a molecular relapse (defined as increase in MRD level by at least 1 log [10-fold] to a level greater than or equal to 5 x 10-4 despite a normal percentage [<5%] of myeloblasts in the bone marrow [BM] aspirate and peripheral blood [PB], and in the absence of proven histological extramedullary relapse). Eligible subjects have a documented diagnosis of AML with at least one of the following molecular aberrations t(8;21), RUNX1-RUNX1T1, inv(16), CBFb/MYH11, t(9;11), MLL-AF9, NPM1 mutation, or FLT3-ITD mutation. Enrolled/randomized pediatric subjects will be followed with regular MRD testing in order to detect a molecular relapse.

In the safety run-in part, up to 12 subjects aged 3 months to less than 18 years will be enrolled. Six subjects will be enrolled in the first cohort of 100 mg/m2 azacitidine administered intravenously (IV) on Days 1 to 7 of a 28-day cycle. Six additional subjects could be enrolled into a second cohort of 75 mg/m2 azacitidine administered IV on Days 1 to 7 of a 28-day cycle depending on the safety and tolerability results of the 100 mg/m2 cohort.

In the randomized part of the study at least 68 subjects will be randomized (or more depending on whether at least 64 subjects are evaluable for the primary endpoint), with at least 60 of the subjects being less than 18 years of age.

Both parts of the study, the safety run-in part and the randomized part, will contain 3 periods: the screening period, the treatment period and the follow-up period. The screening period will last no more than 10 days in the safety run-in part after which the subjects may be enrolled and treated. In the randomized part, the screening period will last an indefinite amount of time until detection of a molecular relapse in the PB followed by confirmation of the relapse in both PB and BM aspirate, at which point the subject may then be randomized. Subjects will be treated with azacitidine (safety run-in part) or in accordance to their assigned treatment arm (randomized part). Upon discontinuation from the treatment period, subjects will enter into the follow-up period which will last up to 2 years from last patient enrolled/randomized.

DETAILED DESCRIPTION:
Study Population Subjects with AML in molecular relapse after CR1, aged 3 months to less than 18 years of age for the safety run-in part, and 3 months to less than 21 years of age for the randomized part.

Length of Study Study duration is estimated to last up to approximately 9 years from the time of the first subject enrollment until completion of the follow-up period for all subjects enrolled/randomized. Estimated duration is based on expected duration of the study treatment/'watch and wait' period (3 months) and completion of the follow-up period (2 years from randomization of last subject).

The End of Trial is defined as either the date of the last visit of the last subject to complete the study, or the date of receipt of the last data point from the last subject that is required for primary, secondary and/or exploratory analysis, as pre-specified in the protocol and/or the Statistical Analysis Plan, whichever is the later date.

Study Treatments Safety Run-in Part Intravenous azacitidine 100 mg/m2 with a possible decrease to a cohort of 75 mg/m2, Days 1 to 7 of a 28-day cycle for a maximum of 3 cycles.

Randomized Part Intravenous azacitidine dose established during the safety run-in part on Days 1 to 7 of a 28-day cycle for a maximum of 3 cycles (for subjects randomized to the azacitidine arm).

Overview of Efficacy Assessments The primary endpoint of the randomized part, PFR at Day 84 (±4 days) post randomization, will be assessed at Day 80 to 88 (approximately end of Cycle 3 of active treatment) post randomization for both the control and the experimental arm. In case of clinical relapse, the investigator will be asked to document it and to evaluate the morphology and immunophenotyping in BM aspirate and PB. This must be done according to standardized diagnostic procedures contained in the AML BFM 2012 guidelines (Creutzig, 2012).

Overview of Safety Assessments Subject safety will be assessed at each visit during the study. Any AE will be reported and recorded in an AE electronic case report form (eCRF). For serious adverse events (SAEs) an expedited reporting procedure will be used in addition to an AE eCRF. The rate of AEs and SAEs, including second malignancies and cardiovascular events which are events of special interest for this study, and abnormal laboratory values and vital signs (NCI CTC Criteria version 4.0 to be used to grade AEs) will be collected while the subject is on study therapy and during the 'watch and wait' period. Once the subject starts the next-line therapy or has a HSCT, only SAEs related to study treatment (experimental arm) or HSCT will be collected for the safety analysis.

Overview of Statistical Methods Subjects from both the safety run-in part and randomization part shall be used for analysis of the safety and efficacy endpoints which are common to both parts of the study. In addition, a PK analysis will be performed on subjects from the safety run-in part, and analysis of the PFR endpoint and all other endpoints unique to the randomized part will only be performed on randomized subjects.

One interim analysis for futility of the primary endpoint is planned during the randomization part of the study once the first 32 (50% of 64) randomized subjects become evaluable for the primaryendpoint analysis. The study will be stopped if the criteria for futility is met.

Subject demographic and baseline characteristics, disposition, and safety data will be presented by study part as well as treatment dose (safety run-in part) and study arm (randomized part) as well as in aggregate for all subjects receiving azacitidine regardless of study part. All efficacy based endpoints will be presented by treatment arm.

First data analysis and reporting of the safety run-in part will be conducted once the final dose assessment SMC meeting has been held (final safety run-in SMC date = data cut-off of initial analysis of safety run-in part). This analysis will consist of the safety run-in primary endpoint and the PK secondary endpoint only. All other safety run-in part secondary endpoints will be analyzed at the time of analysis and reporting of data from the randomized part.

In addition to PK data analysis, all other secondary endpoints can only be analyzed and reported as and when required based on subjects who have had at least 6 months from enrollment (safety run-in part) or randomization (randomization part).

ELIGIBILITY:
Inclusion Criteria:

Safety Run-in Part:

1. Understand and voluntarily provide permission (subjects and when applicable, parental/legal representative(s)) to the informed consent/assent form (ICF/IAF) prior to conducting any study related assessments/procedures.
2. Able to adhere to the study visit schedule and other protocol requirements.
3. Male or Female subjects aged 3 months to less than 18 years old at the time of informed consent/assent.
4. Documented diagnosis of Acute myeloid leukemia (AML) according to World Health Organization (WHO) classification with at least one of the following molecular aberrations below:

   1. t(8;21), RUNX1-RUNX1T1
   2. inv(16), CBFb/MYH11
   3. t(9;11), MLL-AF9
   4. NPM1 mutation
   5. FLT3-ITD mutation.
5. Documentation of molecular remission (MRD less than 5 x 10-4) confirmed at the start of last consolidation course or within 1 month after completion of consolidation treatment.
6. Detection of molecular relapse in the Peripheral Blood (PB) by real-time quantitative polymerase chain reaction (RQ-PCR) within the 7 days prior to signing informed consent/assent form and confirmation of relapse during the screening period. Molecular relapse is defined as an increase in molecular remission (MRD) level of a subject-specific fusion gene or aberration by at least 1 log (10-fold) to a level of at least 5 x 10-4. For subjects who are MRD negative, the rise should be at least 1 log (10-fold) greater than previous sensitivity to a level of 5 x 10-4 or above. An increase in PB must be confirmed in PB and bone marrow (BM) aspirate by RQ-PCR. Confirmation of a molecular relapse is given if the MRD positivity is at the same level or higher in the PB and BM sample compared to the PB MRD levels at the detection of the relapse and in the absence of clinical relapse (defined as at least 5% blasts in PB and/or BM and/or proven histological extramedullary relapse).
7. Lansky play score at least equal to 50; or Karnofsky performance status at least equal to 50, whichever is applicable.
8. Females of Childbearing Potential and male subjects that have reached puberty and are younger than 18 years of age must agree to undergo physician-approved reproductive education and discuss the side effects of the study therapy on reproduction with parent/parents and/or guardian/guardians.
9. Females of Childbearing Potential, defined as females who have achieved menarche and/or 8 years or older and have not undergone a hysterectomy or bilateral oophorectomy, must meet the following conditions below.

   1. Have a negative serum pregnancy test within 72 hours prior to starting study therapy as verified by the study doctor. Agree to ongoing pregnancy testing during the course of the study and after end of study therapy at the 28-day follow-up visit. This applies even if the subject practices true abstinence* from heterosexual contact.
   2. Female subjects must, as appropriate to age and the discretion of the study physician,either commit to true abstinence from heterosexual contact (which must be reviewed on a monthly basis) and/or agree to the use of approved contraceptive method (eg, oral,injectable, or implantable hormonal contraceptive; tubal ligation; intra-uterine device; or vasectomized partner) while on azacitidine; and for 3 months following the last dose.
10. Male subjects must as appropriate to age and the discretion of the study physician:

    1. Agree to use a condom during sexual contact with a pregnant female or a female of childbearing potential while participating in the study, during dose interruptions and for at least 3 months following azacitidine discontinuation, even if he has undergone a successful vasectomy.

Randomized Part (at the time of signing ICF/IAF):

1. Understand and voluntarily provide permission (subjects and when applicable,parental/legal representative(s)) to the ICF/IAF prior to conducting any study related assessments/procedures.
2. Able to adhere to the study visit schedule and other protocol requirements.
3. Male or female subjects aged 3 months to less than 21 years old at the time of informed consent/assent. Note: Minimum of 60 subjects less than 18 years of age must be included. The remainder of the randomized subjects may be greater than or equal to 18 but less than 21 years of age.
4. Documented diagnosis of AML, according to WHO classification with at least one of the following molecular aberrations below that is determined by the central laboratory to be present using BM aspirate from initial diagnosis,:

   1. t(8;21), RUNX1-RUNX1T1
   2. inv(16), CBFb/MYH11
   3. t(9;11), MLL-AF9
   4. NPM1 mutation
   5. FLT3-ITD mutation.
5. Documentation of molecular remission (MRD less than 5 x 10-4) confirmed at the start of last consolidation course or within 1 month after completion of consolidation treatment.

Randomized Part (criteria must be checked at Predrug Verification Visit and re-checked at randomization):

1. Predrug verification visit should occur within 7 days of detection of molecular relapse in the PB by RQ-PCR during the screening period. Molecular relapse is defined as an increase in MRD level of a subject-specific fusion gene or aberration by at least 1 log (10-fold) to a level of at least 5 x 10-4. For subjects who are MRD negative, the rise should be at least 1 log (10-fold) greater than previous sensitivity to a level of 5 x 10-4 or above. An increase in PB must be confirmed in PB and BM aspirate by RQ-PCR. Confirmation of a molecular relapse is given if the MRD positivity is at the same level or higher in the PB and BM sample compared to the PB MRD levels at the detection of the relapse and in the absence of clinical relapse (defined as at least 5% blasts in PB and/or BM and/or proven histological extramedullary relapse).
2. Lansky play score at least equal to 50; or Karnofsky performance status at least equal to 50, whichever is applicable.
3. Females of Childbearing Potential and male subjects that have reached puberty and are:

   1. Younger than 18 years of age must agree to undergo physician-approved reproductive education and discuss the side effects of the study therapy on reproduction with parent/parents and/or guardian/guardians.
   2. Between 18 and 21 years of age must agree to undergo physician-approved reproductive education and discuss the side effects of the study therapy on reproduction with the study physician.
4. Females of Childbearing Potential, defined as females who have achieved menarche and/or 8 years or older and have not undergone a hysterectomy or bilateral oophorectomy, must meet the following conditions below.

   1. Have a negative serum pregnancy test within 72 hours prior to randomization as verified by the study doctor. Agree to ongoing pregnancy testing during the course of the study and after end of study therapy at the 28-day follow-up visit. This applies even if the subject practices true abstinence* from heterosexual contact.
   2. Female subjects must, as appropriate to age and the discretion of the study physician, either commit to true abstinence* from heterosexual contact (which must be reviewed on a monthly basis) and/or agree to the use of approved contraceptive method (eg, oral, injectable, or implantable hormonal contraceptive; tubal ligation; intra-uterine device; or vasectomized partner) while on azacitidine; and for 3 months following the last dose.
5. Male subjects must as appropriate to age and the discretion of the study physician:

   1. Agree to use a condom during sexual contact with a pregnant female or a female of childbearing potential while participating in the study, during dose interruptions and for at least 3 months following azacitidine discontinuation, even if he has undergone a successful vasectomy.

      * True abstinence is acceptable when this is in line with the preferred and usual lifestyle of the subject. [Periodic abstinence (eg, calendar, ovulation, symptothermal, postovulation methods) and withdrawal are not acceptable methods of contraception].

Exclusion Criteria:

Safety Run-in Part (criteria must be checked at Screening and re-checked on Cycle 1 Day

The presence of any of the following will exclude a subject from enrollment:

Concomitant Treatment

1. Concomitant treatment with any other anticancer therapy except those specified in protocol.
2. Received maintenance therapy after end of consolidation therapy and CR1.

   Prior Treatment
3. HSCT (hematopoietic stem cell transplantation) within previous 3 months.
4. Treated by any investigational agent in a clinical study within previous 4 weeks.

   Medical Condition/Laboratory
5. Pregnant or lactating.
6. Symptomatic central nervous system (CNS)-involvement or isolated extramedullary disease at initial diagnosis.
7. FAB (French-American-British) type M3 leukemia (acute promyelocytic leukemia)
8. Therapy-related AML
9. AML of Down syndrome or other congenital syndromes giving rise to leukemia or treatment complications.
10. Symptomatic cardiac disorders (CTCAE (Common Terminology Criteris for Adverse Events) Grade 3 or 4).
11. Evidence of invasive fungal infection or other severe systemic infection requiring treatment doses of systemic/parenteral therapy including known active viral infection with human immunodeficiency virus (HIV) or Hepatitis type B and C.
12. Any other organ dysfunction (NCI CTCAE v4 (National Cancer Institute Common Terminology Criteria for Adverse Events Grade 4) that will interfere with the administration of the therapy according to this protocol.
13. Acute effects of prior chemotherapy/stem cell transplantation.
14. Hypersensitivity to azacitidine.
15. Serum Bilirubin above 1.5 x ULN.
16. Aspartate aminotransferase (AST)/alanine aminotransferase (ALT) above 3 x ULN.
17. Any significant medical condition including the presence of laboratory abnormalities, which places the subject at unacceptable risk if he/she were to participate in the study or that would prevent the subject from participating in the study.

Randomized Part (at the time of signing ICF/IAF):

The presence of any of the following will exclude a subject from enrollment:

Concomitant Treatment

1. Concomitant treatment with any other anti-cancer therapy except those specified in protocol.
2. Received maintenance therapy after end of consolidation therapy and CR1.

   Prior Treatment
3. HSCT within previous 3 months.
4. Treated by any investigational agent in a clinical study within previous 4 weeks.

   Medical Condition/Laboratory
5. Symptomatic CNS-involvement or isolated extramedullary disease at initial diagnosis.
6. FAB type M3 leukemia (acute promyelocytic leukemia)
7. Therapy-related AML
8. AML of Down syndrome or other congenital syndromes giving rise to leukemia or treatment complications.
9. Acute effects of prior chemotherapy/stem cell transplantation.
10. Hypersensitivity to azacitidine.

Randomized Part (criteria must be checked at Predrug Verification Visit and re-checked at randomization):

The presence of any of the following will exclude a subject from randomization:

Prior Treatment

1. Treated by any investigational agent in a clinical study within previous 4 weeks.

   Medical Condition/Laboratory
2. Pregnant or lactating.
3. Symptomatic cardiac disorders (CTCAE Grade 3 or 4).
4. Evidence of invasive fungal infection or other severe systemic infection requiring treatment doses of systemic/parenteral therapy including known active viral infection with human immunodeficiency virus (HIV) or Hepatitis type B and C.
5. Any other organ dysfunction (NCI CTCAE v4.0 Grade 4) that will interfere with the administration of the therapy according to this protocol.
6. Serum bilirubin above 1.5 x ULN.
7. AST/ALT above 3 x ULN.
8. Any significant medical condition including the presence of laboratory abnormalities, which places the subject at unacceptable risk if he/she were to participate in the study or that would prevent the subject from participating in the study.

Ages: 3 Months to 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 7 (Actual)
Dates: Start 2015-08-12 (Actual); Primary Completion 2018-10-10 (Actual); Study Completion 2019-10-08 (Actual)

PRIMARY OUTCOMES:
Adverse Events (AEs) | Up to Day 28
  All reported adverse events during the first treatment cycle
Dose-limiting toxicities (DLTs) | up to Day 28
  Number of participant with DLT
  The rate of the following treatment-related DLTs as per National Cancer Institute Common Terminology Criteria for Adverse Events (NCI CTCAEs) version 4.0, occurring during Cycle 1 only will be considered in determining the tolerability of the 100 mg/m2 dose of azacitidine:
  * Grade 4 nonhematologic toxicity (excluding transient transaminase elevation)
  * Grade 3 nonhematological toxicity lasting more than 7 days despite optimal treatment with standard supportive measures
  * Grade 3 or 4 hematologic toxicity requiring treatment delay greater than 21 days (disease-related Grade 3 or 4 hematologic toxicity will not be counted as a DLT)
Progression-free rate at Day 84 post randomization | up to Day 84
  Proportion of subjects free from clinical progression (clinical relapse and death from any cause) and from molecular progression (defined as lack of stabilization or lack of decrease in molecular aberrations concerning FLT3-ITD mutated, CBF leukemias (eg, t(8;21) and/or inv(16)), MLL-gene rearrangements or NPM1-mutations using central assessment of BM samples by the central laboratories identified for the study, obtained at time points identically prespecified in both randomization arms) at Day 84 (±4 days) post randomization.

SECONDARY OUTCOMES:
Pharmacokinetics - Cmax | Up to Day 7
  Maximum observed concentration in plasma
Pharmacokinetics - Tmax | Up to Day 7
  Observed time to maximum plasma concentration
Pharmacokinetics - AUCt | Up to Day 7
  Area under the plasma concentration-time curve from time zero to the last quantifiable time point
Pharmacokinetics - AUC∞ | Up to Day 7
  Area under the plasma concentration-time curve from time zero to infinity
Pharmacokinetics - λz | Up to Day 7
  Terminal phase rate constant, determined by linear regression of the terminal points of the log-linear plasma concentration-time curve
Pharmacokinetics - t½ | Up to Day 7
  Terminal phase half-life, will be calculated according to the following equation:t½ = 0.693/λz
Pharmacokinetics - CL | Up to Day 7
  Total clearance, calculated as Dose/AUC∞
Pharmacokinetics - Vz | Up to Day 7
  volume of distribution will be calculated according to the equation: Vz = (CL)/λz
Changes in DNA methylation (assessments of BM samples using Nano-HELP assay) | up to Day 60
  Descriptive analyses if the level of DNA methylation at certain CpG loci may predict the response or resistance to azacitidine with regard to the following efficacy endpoints: response, LFS, and OS.
Leukemia-free survival (LFS) | Up to 9 years
  Leukemia-free survival is defined as the time from study enrollment (safety run-in part) or randomization (randomized part) until transition to leukemia progression or death.
Minimal residual disease pre-, and 3 and 6 months post-HSCT | up to 9 years
  Minimal residual disease levels will be assessed across time points
Overall survival | up to 9 years
  Overall survival is the time from study enrollment (safety run-in part) or randomization (randomized part) until death from any cause.
Proportion treated with HSCT | Up to 9 years
  The proportion of subjects undergoing HSCT during the conduct of this study over the total number of subjects enrolled into this study.
Molecular response | up to Day 84
  Molecular response is the number of subjects with molecular response (1 log or more decrease in defined MRD molecular markers from baseline) divided by the number of subjects within the analysis population.
Treatment-related mortality/morbidity | up to 9 years
  All reported SAEs and Deaths during the duration of the study conduct.
Toxicity after HSCT | up to 9 years
  All reported SAEs and deaths post HSCT during the duration of the study conduct
Adverse Events (AEs) | up to 9 years
  All reported adverse events during the duration of the study conduct

CONTACTS AND LOCATIONS:
Overall Officials: Bouchra Benettaib, MD, Study Director — Celgene Corporation
Locations (8):
- Rigshospitalet, Copenhagen, Denmark
- Germany (5):
  - Charite Berlin, Berlin
  - Universitatsklinikum Essen, Essen
  - Klinikum der Johann Wolfgang Goethe-Universität Frankfurt/Main, Frankfurt am Main
  - Universitatsklinik, Freiburg im Breisgau
  - Medical School of Hannover, Hanover
- Netherlands (2):
  - VU University Medical Center, Amsterdam
  - Erasmus University Medical Center, Rotterdam

REFERENCES:
- See also: Expanded Access for CC-486 — https://clinicaltrials.gov/ct2/show/NCT02450877?term=AZA-AML-004&rank=1